CLINICAL TRIAL: NCT03285672
Title: A Phase 2, Randomized, Double-blind, Placebo Controlled, Single Dose-level, Proof-of-concept Study Evaluating FP-101 for the Treatment of Vasomotor Symptoms in Postmenopausal Women
Brief Title: FP-101 for the Treatment of Hot Flashes in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fervent Pharmaceuticals (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FERV001
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2018-10

CONDITIONS: Hot Flashes
Keywords: Hot Flashes, vasomotor symptoms, postmenopausal
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): FP-101
  Interventions: Drug: FP-101
- Arm 2 (Placebo Comparator): Placebo Comparator
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: FP-101 — Dose 1
  Arms: Arm 1
Drug: Placebo Comparator — Dose 1
  Arms: Arm 2

SUMMARY:
The purpose of the study is to determine the efficacy of FP-101 versus placebo for the treatment of hot flashes in postmenopausal women.

DETAILED DESCRIPTION:
Vasomotor symptoms, commonly known as hot flashes or hot flushes, are the most common symptoms experienced by women who are perimenopausal or postmenopausal. FP-101 is postulated to mediate one of the mechanisms thought to drive hot flashes in post-menopausal women. This study will evaluate the efficacy and safety of FP-101 for the treatment of hot flashes in post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be enrolled in the main study only if they meet all of the following criteria:

* Subject must be a female >40 years of age at screening.
* Subject must have reported more than 7 to 8 moderate-to-severe hot flashes per day or 50 to 60 hot flashes per week for at least 30 days prior to the Screening Visit of sufficient severity to cause desire for therapeutic intervention.
* Subject must meet 1 of the following criteria:

  * Spontaneous amenorrhea for at least 12 consecutive months.
  * Amenorrhea for at least 6 months and meet the biochemical criteria for menopause (FSH ≥40 mIU/mL).
  * Bilateral oophorectomy or salpingo-oophorectomy ≥6 weeks prior to enrollment with or without hysterectomy.
* A subject who is not at least 2 years postmenopausal must use adequate nonhormonal contraception (eg, barrier methods such as an intrauterine device, diaphragm, cervical cap, or condom) during study participation.
* Subject must be willing and able to be compliant with the protocol and provide a voluntary written informed consent.

Exclusion Criteria:

* Subject has a history of hypersensitivity or adverse reaction to FP-101 or its excipients
* Subject is a known non-responder to previous SSRI or SNRI treatment for VMS
* Subject has a history of self-injurious behavior.
* Subject has a lifetime history of a clinical diagnosis of major depression or treatment for major depressive disorder.
* Subject has a history of clinical diagnosis of borderline personality disorder.
* Subject has a history of, or is currently presenting with, substance use disorder as defined by the 5th Edition of the Diagnostic and Statistical Manual (DSM-5).
* Subject has a history of psychiatric disorders, including a lifetime history of major depressive disorder, bipolar disorder, panic disorder, generalized anxiety, psychotic disorders, suicidality or suicidal ideation, or post-traumatic stress disorder.
* Subject has a history of hypertension and is not on a stable dose of antihypertensive medications for at least 30 days prior to screening.
* Subject is currently taking MAOIs, thioridazine, or pimozide.
* Subject is currently taking tamoxifen, other selective estrogen receptor modulators, or other hormone deprivation therapy.
* Subject exhibits evidence of impaired liver function upon entry into the study (values ≥2 times the upper limit of normal for aspartate transaminase and/or alanine transaminase, or serum bilirubin ≥1.3 mg/dL) or, in the Investigator's opinion, exhibits liver function impairment to the extent that the subject should not participate in the study.
* Subject has clinically unstable cardiac disease, including unstable atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, or active myocardial ischemia.
* Subject exhibits evidence of impaired kidney function upon entry into the study (i.e., serum creatinine >1.5 mg/dL) or known renal stricture.
* Subject has biliary tract disease, adrenal cortical insufficiency, or any other medical condition that, in the Investigator's opinion, is inadequately treated and precludes entry into the study.
* Subject has thyroid disease, unless subject is clinically stable with normal thyroid indices and is on maintenance thyroid medication (e.g., levothyroxine or liothyronine) for ≥6 months prior to screening.
* Subject exhibits a positive urine pregnancy test result at screening or at any time during study

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 109 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint for the main study is the change in the frequency of moderate-to-severe hot flashes. | Baseline to Week 8

SECONDARY OUTCOMES:
Change in the severity of moderate-to-severe hot flashes. | Baseline to Week 8
Change in the severity of moderate-to-severe hot flashes. | Baseline to Week 4
Change in the frequency of moderate-to-severe hot flashes. | Baseline to Week 4

CONTACTS AND LOCATIONS:
Overall Officials: George Raad, Study Director — PMG Research of Charlotte, LLC
Locations (12):
- United States (12):
  - PMG Research of Christie Clinic, LLC, Champaign, Illinois
  - PMG Research of Cary, LLC, Cary, North Carolina
  - PMG Research of Charlotte, LLC, Charlotte, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Nash OB/GYN, Rocky Mount, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - PMG Research of Charleston, LLC, Mt. Pleasant, South Carolina
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - PMG Research of Knoxville, Oak Ridge, Tennessee

IPD SHARING:
Plan to Share IPD: No